CLINICAL TRIAL: NCT05675904
Title: Textbook Outcome in Colon Carcinoma: Implications for Overall Survival and Disease-free Survival.
Brief Title: Textbook Outcome in Colon Carcinoma
Status: Completed | Type: Observational
Sponsor: Hospital General Universitario de Alicante (Other)
Responsible Party: Principal Investigator, Candido Fernando Alcazar-Lopez, Principal Investigator, Physician, Hospital General Universitario de Alicante
Other Study IDs: 12/2022
Record Dates: First submitted 2022-12-17; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Outcome Assessment; Cancer of Colon
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Yes Textbook Outcome: Patients undergoing scheduled colon cancer surgery with a R0 resection, number of isolated nodes ≥12, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days
  Interventions: Procedure: Colon oncological resection
- No Textbook outcome: Patients undergoing scheduled colon cancer surgery without any of the following items: R0 resection, number of isolated nodes ≥12, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days
  Interventions: Procedure: Colon oncological resection

INTERVENTIONS:
Procedure: Colon oncological resection — Scheduled colon cancer surgery

SUMMARY:
BACKGROUND:

Textbook outcome (TO) is a multidimensional quality management tool that uses a set of traditional surgical measures to reflect an "ideal" surgical result for a particular pathology. The aim of the present study is to record the rate of TO in patients undergoing elective surgery for colon cancer.

MATERIAL AND METHODS:

Retrospective study of all patients undergoing scheduled colon cancer surgery at a Spanish university hospital from September 2012 to August 2016. Patients with rectal cancer were excluded. The variables included in the definition of TO were: R0 resection, number of isolated nodes ≥12, no Clavien-Dindo ≥IIIa complications, no prolonged stay, no readmissions, and no mortality in the first 30 days.

The main objective of this study is to analyse the achievement of TO in a series of patients undergoing scheduled colon cancer resection at the Doctor Balmis General University Hospital in Alicante, Spain. The investigators assess the relationship between TO and overall and disease-free survival, and analyse the indicators included in the definition of TO in colon cancer surgery in order to establish recommendations for its standardization.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective colon cancer resection with confirmed histological diagnosis were eligible for the study

Exclusion Criteria:

* Age under 18 years
* Emergency surgery
* Resections of the rectum or resections for pathologies other than cancer
* Follow-up of less than two years (with the exception of patients who died)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colon cancer resection with confirmed histological diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Textbook Outcome | September 2012- August 2016
  analyse the achievement of Textbook Outcome in a series of patients undergoing scheduled colon cancer resection
Overall survival | From surgery to 160 months
  relationship between Textbook Outcome and overall survival
disease-free survival | From surgery to 160 months
  relationship between Textbook Outcome and disease-free survival

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Dr. Balmis, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No